CLINICAL TRIAL: NCT05193045
Title: Prognosis of Klebsiella ESBL Sepsis: Role of 2-HYDRoxy-myristate in Endotoxin Structure
Acronym: PoKES2_HYDRES
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PoKES2_HYDRES
Record Dates: First submitted 2021-12-31; First posted 2022-01-14 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Klebsiella Infections
MeSH Terms: conditions — Klebsiella Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infections constitute a multiple and heterogeneous set of pathologies, and the first cause of mortality worldwide. Among them, sepsis is a more recent nosological entity, including the most severe forms of acute infectious pathologies, its frequency increasing considerably over time. It is considered to be the cause of more than 27 million deaths per year, more than 4,000 deaths per day in the United States and about 200 deaths per day in intensive care units in France.

The occurrence of hemodynamic failure within visceral damage is a poor prognostic factor, the lethality in this situation can reach 60% of affected patients. The amount of organ dysfunction is also prognostic. More worryingly, the initial mortality is aggravated by the persistence of the negative evolution after hospital treatment, the 5-year prognosis being significantly more severe in the population of patients treated for sepsis than in the general population, particularly in the case of respiratory or cardiovascular damage during the stay in intensive care. The most frequent causes of these severe infections in the ICU are lower respiratory infections, particularly pneumonia acquired under mechanical ventilation, urinary tract infections and digestive tract infections.

Sepsis corresponds to an infection of particular severity, which results in the association of organ failures, the type and severity of which vary according to the patient, the origin of the infection and the pathogen responsible. The severity of the picture will require specific management and may necessitate the introduction of organ supplements or even lead to death in the most serious forms.

Infections by enterobacteria and in particular Klebsiella spp. are frequent in the intensive care unit. The association with antibiotic resistance and especially with ESBL production is a daily clinical situation. During these infections, the prognosis is variable, sometimes very poor, without it being possible to determine whether this evolution is due to antibiotic resistance or to the virulence of the pathogen. The objective of this work is to study the structure of lipid A of ESBL-producing Klebsiella strains responsible for nosocomial infections. This study is part of the "EVENT" protocols of which it is an ancillary analysis.

The objective of this study is to evaluate the role of the presence of 2-hydroxymyristate within lipid A of the lipopolysaccharide in the prognosis of ESBL-producing Klebsiella infections in the ICU. The secondary objectives correspond to the evaluation of the vital prognosis according to the infected organ (lung, kidney, digestive system), and the presence of 2-hydroxymyristate and the risk of bacteremia.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patient hospitalized in an intensive care unit
* Patient with a nosocomial infection with ESBL-producing Klebsiella
* French-speaking patient

Exclusion Criteria:

* Patient with a severe psychiatric disorder
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient who objects to the use of his or her data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These patients were hospitalized in the ICU with nosocomial ESBL-producing Klebsiella infection between 2011 and 2016.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2021-11-28 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Role of 2-hydroxymyristate within lipid A of lipopolysaccharide in the prognosis of ESBL-producing Klebsiella infections in the ICU | Day 128
  This outcome corresponds to the mortality in intensive care.

SECONDARY OUTCOMES:
Evaluation of the vital prognosis according to the infected organ (lung, kidney, digestive system) at day 28 | Day 28
  This outcome corresponds to the mortality rate at day 28.
Evaluation of the vital prognosis according to the infected organ (lung, kidney, digestive system) at 3 months. | Month 3
  This outcome corresponds to the mortality rate at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Francois PHILIPPART, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Prescott HC, Angus DC. Enhancing Recovery From Sepsis: A Review. JAMA. 2018 Jan 2;319(1):62-75. doi: 10.1001/jama.2017.17687. PMID 29297082
- [Background] Brun-Buisson C, Meshaka P, Pinton P, Vallet B; EPISEPSIS Study Group. EPISEPSIS: a reappraisal of the epidemiology and outcome of severe sepsis in French intensive care units. Intensive Care Med. 2004 Apr;30(4):580-8. doi: 10.1007/s00134-003-2121-4. Epub 2004 Mar 2. PMID 14997295
- [Background] de Grooth HJ, Postema J, Loer SA, Parienti JJ, Oudemans-van Straaten HM, Girbes AR. Unexplained mortality differences between septic shock trials: a systematic analysis of population characteristics and control-group mortality rates. Intensive Care Med. 2018 Mar;44(3):311-322. doi: 10.1007/s00134-018-5134-8. Epub 2018 Mar 15. PMID 29546535
- [Background] Rhee C, Dantes R, Epstein L, Murphy DJ, Seymour CW, Iwashyna TJ, Kadri SS, Angus DC, Danner RL, Fiore AE, Jernigan JA, Martin GS, Septimus E, Warren DK, Karcz A, Chan C, Menchaca JT, Wang R, Gruber S, Klompas M; CDC Prevention Epicenter Program. Incidence and Trends of Sepsis in US Hospitals Using Clinical vs Claims Data, 2009-2014. JAMA. 2017 Oct 3;318(13):1241-1249. doi: 10.1001/jama.2017.13836. PMID 28903154
- [Background] Shankar-Hari M, Harrison DA, Ferrando-Vivas P, Rubenfeld GD, Rowan K. Risk Factors at Index Hospitalization Associated With Longer-term Mortality in Adult Sepsis Survivors. JAMA Netw Open. 2019 May 3;2(5):e194900. doi: 10.1001/jamanetworkopen.2019.4900. PMID 31150081
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Crit Care Med. 2017 Mar;45(3):486-552. doi: 10.1097/CCM.0000000000002255. PMID 28098591